CLINICAL TRIAL: NCT03484741
Title: A Preliminary Safety and Efficacy Evaluation of Mesenchymal Stem Cell Transplantation for Type 1 Diabetes Mellitus (T1DM) Patients
Brief Title: Mesenchymal Stem Cell Therapy for Type 1 Diabetes Mellitus Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Van Hanh General Hospital (Other)
Collaborators: University of Science Ho Chi Minh City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIME 1001; DIME 1001 (Other: Ministry of Health, Viet Nam)
Record Dates: First submitted 2018-03-16; First posted 2018-04-02 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC and PRP (Experimental): 15 patients will be given autologous bone marrow-derived mesenchymal stem cells (BM-MSC) and mesenchymal stem cell from allogeneic umbilical cord tissue (UC-MSC) combined with platelet-rich plasma (PRP) by intravenous infusion.
  Interventions: Biological: MSC and PRP

INTERVENTIONS:
Biological: MSC and PRP — MSC are collected from autologous bone marrow mononuclear cells (BMNC) and allogeneic umbilical cord tissue (UC-MSC) under sterile conditions and combined with activated platelet-rich plasma (PRP) to treat this disease.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of mesenchymal stem cells (MSCs) transplantation for type 1 Diabetes Mellitus patients.

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSCs) are collected from autologous bone marrow mononuclear cells and allogeneic umbilical cord tissue (UC-MSC).

15 patients with type 1 Diabetes Mellitus will be enrolled and will receive MSCs by intravenous infusion. They were followed up for 6 months after transplantation.

Safety is to assess the occurrence of adverse events (AEs) during either stem cells infusion or by physician assessments.

The primary endpoint is to assess the improvement of patients' Fasting blood glucose, HbA1C, C-peptide, and blood insulin level.

ELIGIBILITY:
Inclusion Criteria:

* Who is diagnosed with Type 1 Diabetes Mellitus according to the ADA, the patients meet at least one of the following criteria:

  * At least one autoantibody associated with Type 1 Diabetes Mellitus such as ICA or GAD.
  * Previously diagnosed at a medical facility with Type 1 Diabetes.
  * Having evidence of insulin depletion based on the test results during screening.
* Patients treated with fixed insulin dose for at least 3 months.
* Males and females between age 18 and 45 years at the screening.
* Patients able to read, write and understand ICF form

Exclusion Criteria:

* Uncontrolled blood pressure at the time of enrollment: systolic pressure >160 mmHg and/or diastolic blood pressure > 100 mmHg.
* Having evidence related to renal dysfunction:

  * creatinine > 1.5 mg/dl or (>133 mmol/L) for men.
  * creatinine > 1.4 mg/dl or (>124 mmol/L) for woman.
  * eGRF < 40 ml/ min
* Proteinuria > 300 mg/day
* Having evidence of ketoacidosis at the time of selection.
* Having evidence of ongoing or frequent hypoglycemia.
* Having severe infection
* Infected with hepatitis B virus or hepatitis C or tuberculosis. Positive results of HbsAg or Anti HCV or/and PCR tuberculosis are only acceptable in case of vaccination and without suspicious signs. All other cases are not accepted even in the absence of clinical signs.
* Diseases detected before/during screening such as cardiovascular disease, respiratory disease ( pulmonary, fibrosis, chronic respiratory failure), liver disease, cancer, neurology, metabolism.
* Having abnormalities in red blood cells such as sickle cells disease.
* Using alcohol and/or tobacco.
* Blood clotting disorders (INR > 1.5, PTT >40, PT > 15).
* Taking any anticoagulant.
* Taking systemic steroids.
* Participate in another clinical study involving experimenting drugs and/or medical equipment.
* Patients who are unable to perform the tests and assessments needed for the study (eg, patients who are unable to perform bone marrow transplantation) or patients who do not agree to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose | every month in the course of 6 months
  Assess the changes in fasting blood glucose level after transplantation
Hemoglobin A1c (HbA1c) level | 1 month, 3 months and 6 months after transplantation
  Assess the changes in HbA1C level after transplantation
Adverse events | during the course of 6 months
  Evaluate the safety of therapy by number record of adverse events (AEs)

SECONDARY OUTCOMES:
Insulin dose | during the course of 6 months
  Reduction of insulin dose after transplantation
C-peptide | every month in the course of 6 months
  Assess the improvement in C-peptide level after transplantation
Blood insulin level | every month in the course of 6 months
  Assess the changes in blood insulin level after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Phuong Le, MSc-MD, Principal Investigator — Stem Cell Unit, Van Hanh General Hospital; Ngoc Phan, MSc, Principal Investigator — Stem Cell Institute, University of Science Ho Chi Minh City
Locations (1):
- Van Hanh Geral Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 6 months after publication
Access Criteria: Type 1 Diabetes Mellitus